CLINICAL TRIAL: NCT04036266
Title: Effect of Medial Open Wedge High Tibial Osteotomy on Clinical and Radiographic Outcomes of Patients With Knee Osteoarthritis : A Retrospective Study
Brief Title: Clinical and Radiographic Outcomes of Medial Open-wedge High Tibial Osteotomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Salah Abdelhamid Ahmed, Resident in orthopedic and traumatology department, Assiut University
Other Study IDs: MOWHTO in OA
Record Dates: First submitted 2019-03-29; First posted 2019-07-29 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: medial open wedge high tibial osteotomy — opening of medial aspects of the proximal tibial metaphysis and change the coronal alignment of the tibia in order to shift the center of force passing axially through the knee from the arthritic region of the knee towards the unaffected side then fixation with a plate (the standard plate is the T-locked plate )

SUMMARY:
Osteoarthritis is a common degenerative disorder of the articular cartilage . Risk factors include genetics, female sex, past trauma, advancing age, and obesity. The diagnosis is based on a history of joint pain worsened by movement, which can lead to disability in activities of daily living .

Diagnosis of knee osteoarthritis can be confirmed based on clinical and/or radiological features. The potential of a progressive disease can be prevented or decreased by earlier recognition and correction of associated factors. Obesity and alignment especially varus malalignment are recognized factors of a progressive disease.

High tibial osteotomy (HTO) is a widely performed procedure, and good results can be achieved with appropriate patient selection and precise surgical technique. It is reported to be an effective treatment for varus knee osteoarthritis (OA) by redistributing the load line within the knee joint . With an HTO, the surgeon aims to change the coronal alignment of the leg in order to shift the center of force passing axially through the knee from the arthritic region of the knee towards the unaffected side. The amount of alignment correction to be performed is calculated before surgery based on the extent of knee arthrosis and on the alignment of the patient's lower limbs on long-leg weight bearing radiographs .

Our study is focused on effectiveness of open wedge High tibial osteotomy on clinical and radiographic outcomes of patients with medial knee osteoarthritis.

DETAILED DESCRIPTION:
The investigators will conduct a retrospective case-series study of at least 40 patients , who underwent medial open-wedge HTO for treatment of medial knee osteoarthritis between January 2016 and January 2019 in our Arthroscopy and Sports Injuries Unit in Orthopaedics Department of Assiut University. Inclusion criteria is Kellgren-Lawrence classification grades 1 to 3; symptomatic unicompartmental osteoarthritis

Pre-operative :

assessment of patients is done clinically using Knee society score (KSS) and visual analogue scale (VAS) (0 mm, no pain;100 mm, worst pain) and radiographic assessment according to Kellgren and Lawrence using anteroposterior (AP) and lateral x-ray views of the knee , a two-leg long standing view with or without slight flexion assessing Femoral-tibial angle (FTA) .

Intra-operative :

After anaesthesia is induced, an arthroscopic examination is performed to define the status of the menisci (excluding significant damage of the lateral compartment), cruciate ligaments, and articular cartilage. meniscal surgery (partial menisectomy/meniscal repair) is performed when necessary, then The medial open wedge high tibial osteotomy (MOWHTO) is performed.

Post-operative :

follow up after at least 1 year post-operative clinically using knee society score (KSS) , visual analogue scale (VAS),Knee Injury and Osteoarthritis Outcome Score(KOOS) , Western Ontario and McMaster Universities Osteoarthritis (WOMAC) index scores and radiological assessment using Anteroposterior and lateral views xrays assessing union two-leg long standing view x ray with or without slight flexion assessing Femoral-tibial angle (FTA) and joint line .

ELIGIBILITY:
Inclusion Criteria:

* Age above 30 years old.
* Patients who had MOWHTO for knee OA within the past 5 years .
* No response to non-surgical treatment (medical and physiotherapy) pre operatively for at least 3 months.
* Intact cruciate ligaments, and Collateral ligaments.

Exclusion Criteria:

* Age less than 30 years old.
* Patients who had HTO for another reasons other than knee OA.
* Combined injury to (collateral ligaments, cruciate ligament).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients older than 30 years old that underwent medial open wedge high tibial osteotomy due to medial osteoarthritis of the knee
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
pain relief is being assessed using Visual analogue scale (VAS) | 1 year up to 5 years post operative
  assessment is done using Visual analogue scale (VAS)

SECONDARY OUTCOMES:
varus malalignment correction of the knee | 1 year up to 5 years post operative
  this is measured using femoral tibial angle

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M. Abdelhamid, PHD, Study Chair — Professor of Orthopedics and Traumatology; Islam K. Ramadan, PHD, Study Director — Lecturer of Orthopedics and Traumatology

REFERENCES:
- [Background] Heidari B. Knee osteoarthritis diagnosis, treatment and associated factors of progression: part II. Caspian J Intern Med. 2011 Summer;2(3):249-55. PMID 24049581
- [Background] Kim YS, Koh YG. Comparative Matched-Pair Analysis of Open-Wedge High Tibial Osteotomy With Versus Without an Injection of Adipose-Derived Mesenchymal Stem Cells for Varus Knee Osteoarthritis: Clinical and Second-Look Arthroscopic Results. Am J Sports Med. 2018 Sep;46(11):2669-2677. doi: 10.1177/0363546518785973. Epub 2018 Aug 6. PMID 30080423
- [Background] Mukherjee K, Latif A, Ranjan AK, Dugar N. High tibial osteotomy--an effective treatment option for osteo-arthritis. J Indian Med Assoc. 2013 Dec;111(12):801-3. PMID 25154146
- [Background] Sinusas K. Osteoarthritis: diagnosis and treatment. Am Fam Physician. 2012 Jan 1;85(1):49-56. PMID 22230308
- [Background] Altay MA, Erturk C, Altay N, Mercan AS, Sipahioglu S, Kalender AM, Isikan UE. Clinical and radiographic outcomes of medial open-wedge high tibial osteotomy with Anthony-K plate: prospective minimum five year follow-up data. Int Orthop. 2016 Jul;40(7):1447-54. doi: 10.1007/s00264-015-2919-z. Epub 2015 Jul 21. PMID 26194919